CLINICAL TRIAL: NCT01405040
Title: Clinical Evaluation of a New Transpulmonary Thermodilution Method to Assess TPTD, GEDV and EVLW
Brief Title: Clinical Evaluation of a New Transpulmonary Thermodilution Method to Assess Thermodilution Cardiac Output, Global End Diastolic Volume and Extravascular Lung Water
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: MIM-0906-0001
Record Dates: First submitted 2011-07-20; First posted 2011-07-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Cardiac Output and Preload Assessment; Lung Water Assessment
Keywords: Cardiac; Output; Preload; Lung; Water

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EV1000 Observational Group: Patient must have an indwelling femoral arterial catheter and central venous catheter considered necessary for routine clinical monitoring; Patient, or legal guardian, will give consent prior to study enrollment and data capture; Patient must be at least 18 years old; Patient height and weight are available prior to study.

SUMMARY:
The primary objective of this study is to obtain the TPTD, GEDV and EVLW measurements from existing indwelling femoral arterial Volume View™ catheter and central venous catheters.

DETAILED DESCRIPTION:
Transpulmonary thermodilution has been proposed to measure transpulmonary thermodilution cardiac output (TPTD), preload (GEDV, global end diastolic volume) and to quantify pulmonary edema (EVLW, extravascular lung water). The method currently available on the market is based on the estimation of time characteristics of the curve (mean transit time and down slope time).

The purpose of this study is to evaluate a new transpulmonary thermodilution method to assess the TPTD, EVLW and GEDV in patients requiring cardiac preload and lung water assessment. Up to one hundred (100) patients will be enrolled at four (4) study sites, (up to 25 subjects at each site). Hôpitaux Universitaires de Genève, Universität Bonn, Stadtspital Triemli Zürich, and Universitätsklinikum Aachen will participate in the study.

This is a prospective, observational data collection study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have clinical need for an indwelling femoral arterial catheter and central venous catheter.
2. Patient, or legal guardian, must sign consent to be in the study prior to data capture.
3. Patient must be at least 18 years old.
4. Patient height and weight are available prior to study.

Exclusion Criteria:

1. Patients with significant aortic valve regurgitation.
2. Patients being treated with an intra-aortic balloon pump.
3. Patients less than 40 kg in weight.
4. Female patients with a known pregnancy or planned pregnancy.
5. Patient is currently participating in an investigational drug or another device study that clinically interferes with the study endpoints.
6. Patients with peripheral vascular disease.
7. Patients with aortic aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all ICU patients requiring cardiac preload and lung water assessment.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
TPTD, GEDV and EVLW measurements to evaluate the precision and accuracy of a novel algorithm in comparison to the widely accepted TPTD method | Up to 72 hours of femoral arterial catheter dwell time.
  This is not an outcome study. This is an observational Study to obtain TPTD, GEDV and EVLW data to evaluate the precision and accuracy of a novel algorithm in comparison to the widely accepted TPTD method using an approach defined by Bland-Altman.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Deyette, RN, CCRP, Study Director — Edwards Lifesciences LLC
Locations (4):
- Germany (2):
  - Universitätsklinikum der RWTH Aachen, Aachen, Pauwelsstrasse 30
  - Der Rheinischen Friedrich-Wilhelms-Universität Bonn, Bonn, Sigmund Freud Strasse 25
- Switzerland (2):
  - Stadtspital Triemli Zürich, Zurich, Birmensdorferstr 497
  - HUG-Hôpitaux Universitalres de Genève, Geneva, Canton of Geneva

REFERENCES:
- [Derived] Bendjelid K, Marx G, Kiefer N, Simon TP, Geisen M, Hoeft A, Siegenthaler N, Hofer CK. Performance of a new pulse contour method for continuous cardiac output monitoring: validation in critically ill patients. Br J Anaesth. 2013 Oct;111(4):573-9. doi: 10.1093/bja/aet116. Epub 2013 Apr 26. PMID 23625132
- [Derived] Kiefer N, Hofer CK, Marx G, Geisen M, Giraud R, Siegenthaler N, Hoeft A, Bendjelid K, Rex S. Clinical validation of a new thermodilution system for the assessment of cardiac output and volumetric parameters. Crit Care. 2012 May 30;16(3):R98. doi: 10.1186/cc11366. PMID 22647561